CLINICAL TRIAL: NCT02532582
Title: Effort to Reduce Postoperative Brachial Neuropraxia Through Nerve Compression
Brief Title: Assessment of Patient Positioning
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Daniela Ladner, Associate Professor of Surgery, Northwestern University
Other Study IDs: STU00105002
Record Dates: First submitted 2015-08-10; First posted 2015-08-26 (Estimated); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Neuropraxia
Keywords: nerve compression
MeSH Terms: conditions — Neuroma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Living Liver Donor Transplant Donors: All adult living liver donors and liver surgery patients at Northwestern Memorial Hospital (same surgical setup is used for living liver donor surgery and liver surgery (e.g. retractors, arterial line for monitoring, surgeons). Living liver donors and liver surgery patients for enrollment to receive neuromuscular monitoring)

SUMMARY:
The purpose of this study is to ultimately prevent injuries to nerves during surgical procedures. Living donor liver transplant or hepatectomy (removal of a piece of the liver) patients will receive an arterial line as standard of care. The arterial line helps monitor blood pressure along with the compression of important vessels during surgery. In addition, research participants will undergo neuromuscular monitoring using Somato-Sensory Evoked Potential (SSEP) or Evoked Potential Assessment Device (EPAD). During an operation, neuromuscular monitoring can tell doctors if the nerves being studied are working normally or if they are at risk for injury. This study will help investigators to understand what kind of monitoring is best to prevent nerve injuries during a surgical procedure.

DETAILED DESCRIPTION:
As standard of care, research participants undergoing a living donor liver transplant or other liver surgeries will receive a right-sided radial arterial line to monitor his/her blood pressure along with the compression of important vessels during surgery. These measurements will be captured throughout the surgical procedure. If blunting of the arterial line wave form occurs, the anesthesiology team alerts the surgical team to release the retractors until the wave form returns to baseline. Depression of the radial arterial line wave form will be captured, time-stamped, and stored by the research transplant anesthesiology team.

Additionally as part of research, participants will receive neuromuscular monitoring using SSEP or EPAD to measure their nerve signals during the surgery (3-6 hours). SSEP or EPAD measurements will occur at the median and ulnar nerve and will be captured throughout the surgical procedure. The research neuromonitoring team will consists of highly skilled technicians, who monitor patients during neurosurgical and orthopedic surgeries. SSEP or EPAD output captured during the surgery will be time-stamped, stored, and interpreted by a Neurologist. To investigate if a correlation exists, SSEP or EPAD abnormalities will be correlated and analyzed with the arterial wave form depressions.

To determine whether a correlation exists with clinical outcomes, a prospective medical record review will be conducted. Before performing the prospective medical record review, authorized research personnel will obtain informed consent from each participant.

ELIGIBILITY:
Inclusion Criteria:

* All adult living liver donors and liver surgery patients at Northwestern Memorial Hospital (surgical setup is similar for living liver donor surgery and liver surgery (e.g. retractors, arterial line for monitoring, surgeons). Investigators will approach both living liver donors and liver surgery patients for enrollment to receive additional neuromuscular monitoring.
* All subjects must have given signed, informed consent prior to registration on the study.

Exclusion Criteria:

* Anyone not meeting the inclusion criteria.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adult living liver donors and liver surgery patients at Northwestern Memorial Hospital (surgical setup is similar for living liver donor surgery and liver surgery (e.g. retractors, arterial line for monitoring, surgeons). Investigators will approach both living liver donors and liver surgery patients for enrollment to receive additional neuromuscular monitoring.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2015-05; Primary Completion 2020-05 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
A change in arterial line wave form and a change in the neuromuscular signal using SSEP or EPAD will be measured and tested with the Pearson correlation coefficient as well as nonparametric Spearman's rank correlation coefficient. | 12 mos
  To establish the correlation between the wave form of the arterial line readings and neuromuscular monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela P Ladner, MD, MPH, Principal Investigator — Northwestern University